CLINICAL TRIAL: NCT03142841
Title: Spanish Online & Telephone Intervention for Caregivers of Veterans With Stroke
Brief Title: Spanish Intervention for Caregivers of Veterans With Stroke
Acronym: RESCUE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IIR 15-117
Record Dates: First submitted 2017-05-01; First posted 2017-05-05 (Actual); Results first posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Depression
Keywords: Depression; Burden; Problem Solving Ability; Caregivers; Stroke; Veterans
MeSH Terms: conditions — Depression; Stroke

STUDY DESIGN:
Intervention Model Description: A two-arm (8-session intervention vs. standard care), randomized controlled clinical trial with three assessment points will be conducted. Baseline measurements will be conducted with the caregivers prior to the intervention. Post-test assessments will be collected at 1 and 12 weeks post-intervention. In addition, the investigators will obtain pre- and post-test measures of Veteran-related variables via CPRS electronic health records. Qualitative interviews will be conducted to assess caregivers' perceptions of the intervention.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The PI and data collectors will be blinded in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Care (No Intervention): The standard care group will receive the usual standard care they would receive had they not been enrolled in this study
- Problem Solving Intervention (Experimental): Participants in the intervention group received an 8-week problem-solving session conducted over the phone by a trainer interventionist. The intervention consists of four components: 1. Introduction to the RESCUE website and the problem-solving method; 2. Illustrative example on how to use the problem-solving approach and the RESCUE website to address caregiving problems; 3. Individualized practice exercise to develop a personalized problem-solving plan; and 4. Summary of the problem-solving method.
  Interventions: Other: RESCUE Problem Solving Intervention

INTERVENTIONS:
Other: RESCUE Problem Solving Intervention — The RESCUE Problem Solving Intervention: This is an education and support intervention for caregivers of Veterans with stroke. The investigators taught study participants the COPE (Creativity, Optimism, Planning, Expert Advice) model of problem solving and guided them through the application of this model in their caregiver role. They also receive tailored stroke education, specific to their needs.
  Arms: Problem Solving Intervention

SUMMARY:
This research study will test a problem-solving intervention for Spanish-speaking stroke caregivers that will be delivered over the telephone and online via the previously developed and nationally available Spanish version of the RESCUE website. The investigators will adapt their previously pilot-tested problem-solving intervention and make it culturally-relevant for Hispanic caregivers. The investigators' main goal is to test the efficacy of a brief, telephone and online problem-solving intervention. The objectives are: 1) reduce caregiver burden and depression, 2) improve caregivers' problem-solving abilities, self-efficacy, and quality of life, 3) improve Veterans' functional abilities and determine the intervention's impact on Veterans' healthcare utilization, 4) determine budgetary impact, and 5) determine caregivers' perceptions of the intervention.

DETAILED DESCRIPTION:
This research study will test a problem-solving intervention for Spanish-speaking stroke caregivers that will be delivered over the telephone and online via the previously developed and nationally available Spanish version of the RESCUE website. The investigators will adapt their previously pilot-tested problem-solving intervention and make it culturally-relevant for Hispanic caregivers. The investigators' main goal is to test the efficacy of a brief, telephone and online problem-solving intervention. The objectives are: 1) reduce caregiver burden and depression, 2) improve caregivers' problem-solving abilities, self-efficacy, and quality of life, 3) improve Veterans' functional abilities and determine the intervention's impact on Veterans' healthcare utilization, 4) determine budgetary impact, and 5) determine caregivers' perceptions of the intervention.

The investigators will conduct a two-arm (8-session intervention vs. standard care), , randomized controlled trial to test a problem-solving intervention for Spanish-speaking stroke caregivers that will be delivered over the telephone and online via the previously developed and nationally available Spanish version of the RESCUE website. A sample of 290 stroke caregivers will be randomly assigned to either an intervention or a standard care group. Eligibility criteria: Hispanic caregivers of Veterans with a primary diagnosis of stroke are eligible for participation if they meet the following criteria: 1) are the primary caregiver and provide the majority of care for a Veteran who has a diagnosis of stroke (ICD9 codes for stroke: 430-438 or ICD 10 codes 160.0 through 169.998) within the last year and who has at least two activity of daily living (ADL) deficits or a new or worsening neurological problem, 2) have Internet access and ability, (either themselves or via a relative or friend) 3) are reachable by cell or home phone, 4) Spanish is their preferred language, 5) have moderate to severe stress, and 6) ) identify self as Hispanic, and 7) agree to random assignment to the intervention or standard care group. We will determine caregiver status.

Baseline measurements will be conducted with the caregivers prior to the intervention. Post-test assessments will be collected at 1 and 12 weeks post-intervention. In addition, the investigators will obtain pre- and post-test measures of Veteran-related variables via Computerized Patient Record System (CPRS) electronic health records. Qualitative interviews will be conducted to assess caregivers' perceptions of the intervention. A general linear mixed model for repeated measures will be used to examine the relationship between treatment assignment and each outcome over time. The investigators will measure the budgetary impact of providing intervention by comparing the costs of the intervention group to the costs of the control group.

ELIGIBILITY:
Inclusion Criteria: Hispanic caregivers of Veterans with a primary diagnosis of stroke are eligible for participation if they meet the following criteria: 1) are the primary caregiver and provide the majority of care for a Veteran who has a diagnosis of stroke (ICD9 codes for stroke: 430-438 or ICD 10 codes 160.0 through 169.998) within the last year and who has at least two activity of daily living (ADL) deficits or a new or worsening neurological problem, 2) have Internet access and ability, (either themselves or via a relative or friend) 3) are reachable by cell or home phone, 4) Spanish is their preferred language, 5) have moderate to severe stress, and 6) ) identify self as Hispanic, and 7) agree to random assignment to the intervention or standard care group.

Random assignment to the intervention or standard care group. The investigators will determine caregiver status.

Exclusion Criteria: The investigators will exclude caregivers who fail to meet one or more of the inclusion criteria or are managing end-of-life issues (stroke survivors are likely to die within five months following discharge).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2024-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivette M Freytes, PhD MEd BA, Principal Investigator — North Florida/South Georgia Veterans Health System, Gainesville, FL
Locations (4):
- United States (3):
  - North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida
  - Orlando VA Medical Center, Orlando, FL, Orlando, Florida
  - James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida
- VA Caribbean Healthcare System, San Juan, PR, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Freytes IM, Schmitzberger MK, Rivera-Rivera N, Lopez J, Motta-Valencia K, Wu SS, Orozco T, Hale-Gallardo J, Eliazar-Macke N, LeLaurin JH, Uphold CR. Study protocol of a telephone problem-solving intervention for Spanish-speaking caregivers of veterans post-stroke: an 8-session investigator-blinded, two-arm parallel (intervention vs usual care), randomized clinical trial. BMC Prim Care. 2023 Mar 17;24(1):73. doi: 10.1186/s12875-022-01929-y. PMID 36932321
- [Background] Freytes IM, Schmitzberger M, Rivera-Rivera N, Lopez J, Mylott D, Motta-Valencia K, Uphold CR. Serving Underserved Veterans and Their Caregiver: Developing Tailored Culturally Relevant Interventions. [Abstract]. Innovation in aging. 2019 Nov 8; 3(Supp 1):S674.
- See also: Testing the Impact of a Spanish Online and Telephone Intervention for Hispanic Caregivers of Veterans with Stroke — https://www.hsrd.research.va.gov/publications/forum/spring23/default.cfm?ForumMenu=spring23-5

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Care Group: The standard care group will receive the usual standard care they would receive had they not been enrolled in this study.
- Intervention Group: Participants in the intervention group received an 8-week problem-solving session conducted over the phone by a trained interventionist. The intervention consists of four components: 1. Introduction to the RESCUE website and the problem-solving method; 2. Illustrative example on how to use the problem-solving approach and the RESCUE website to address caregiving problems; 3. Individualized practice exercise to develop a personalized problem-solving plan; and 4. Summary of the problem-solving method.
  The RESCUE Problem Solving Intervention: This is an education and support intervention for caregivers of Veterans with stroke. The interventionists taught study participants the COPE (Creativity, Optimism, Planning, Expert Advice) model of problem solving and guided them through the application of this model in their caregiver role. Caregivers also received tailored stroke education specific to their needs from the RESCUE website.
Period: Overall Study
Arm/Group | Standard Care Group | Intervention Group
Started | 105 | 105
Completed | 86 | 70
Not Completed | 19 | 35

BASELINE CHARACTERISTICS:
Groups:
- Intervention Group: Participants in the intervention group received an 8-week problem-solving session conducted over the phone by a trainer interventionist. The intervention consists of four components: 1. Introduction to the RESCUE website and the problem-solving method; 2. Illustrative example on how to use the problem-solving approach and the RESCUE website to address caregiving problems; 3. Individualized practice exercise to develop a personalized problem-solving plan; and 4. Summary of the problem-solving method.
  The RESCUE Problem Solving Intervention: This is an education and support intervention for caregivers of Veterans with stroke. The investigators taught study participants the COPE (Creativity, Optimism, Planning, Expert Advice) model of problem solving and guided them through the application of this model in their caregiver role. They also receive tailored stroke education, specific to their needs.
- Total: Total of all reporting groups
Arm/Group | Standard Care Group | Intervention Group | Total
Number analyzed (Participants) | 105 | 105 | 210
Age, Customized [Count of Participants; unit: Participants]
  18 years or older | 105 | 105 | 210
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 92 | 185
  Male | 12 | 13 | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 50 | 51 | 101
  Black | 5 | 13 | 18
  Multi-Racial | 34 | 27 | 61
  Pacific Island Native | 2 | 0 | 2
  Other | 5 | 6 | 11
  Unknown | 9 | 8 | 17
Caregiver- Marital Status [Count of Participants; unit: Participants]
  Single | 11 | 22 | 33
  Married | 74 | 62 | 136
  Living Together with Partner | 8 | 6 | 14
  Divorced or Separated | 11 | 13 | 24
  Widowed | 1 | 1 | 2
  Unknown | 0 | 1 | 1
Caregiver- Education [Count of Participants; unit: Participants]
  Some High School | 5 | 7 | 12
  High School Graduate | 11 | 17 | 28
  Some College/Vocational | 28 | 39 | 67
  College Degree | 43 | 29 | 72
  Masters Degree | 14 | 10 | 24
  Doctoral Degree | 3 | 3 | 6
  Not Answered | 1 | 0 | 1
Caregiver- Income [Count of Participants; unit: Participants]
  < $10,000 per year | 11 | 10 | 21
  $10,000 - $20,000 per year | 24 | 36 | 60
  $20,001 - $30,000 per year | 18 | 19 | 37
  $30,001 - $40,000 per year | 14 | 10 | 24
  $40,001 - $50,000 per year | 16 | 14 | 30
  > $50,000 per year | 20 | 14 | 34
  Unknown | 2 | 2 | 4
Caregiver- Relationship to Veteran [Count of Participants; unit: Participants]
  Spouse | 52 | 44 | 96
  Child | 35 | 35 | 70
  Partner | 5 | 6 | 11
  Parent | 1 | 1 | 2
  Sibling | 2 | 7 | 9
  Other Family Member | 7 | 8 | 15
  Other Type of Relationship | 3 | 4 | 7
Caregiver- Employment [Count of Participants; unit: Participants]
  Full-Time | 27 | 15 | 42
  Part-Time | 8 | 10 | 18
  Retired | 36 | 43 | 79
  Unemployed | 33 | 35 | 68
  Unknown | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Caregiver Depression at 9 Weeks
Description: Caregiver depression as measured by the Center for Epidemiologic Studies Depression-20. The CES-D is a 20 item, four point Likert scale ranging from never (0) to most of the time (3). The minimum value is 0 and the maximum value is 60. The higher score means a worse outcome (more depressed). This tool has good reliability and validity.
Time Frame: 9 weeks after baseline
Population: Data collected from 156 participants who completed the study. Data from caregivers who ended up not meeting study criteria were not included in the analysis of data.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Intervention Group: Participants in the intervention group received an 8-week problem-solving session conducted over the phone by a trained interventionist. The intervention consists of four components: 1. Introduction to the RESCUE website and the problem-solving method; 2. Illustrative example on how to use the problem-solving approach and the RESCUE website to address caregiving problems; 3. Individualized practice exercise to develop a personalized problem-solving plan; and 4. Summary of the problem-solving method.
  The RESCUE Problem Solving Intervention: This is an education and support intervention for caregivers of Veterans with stroke. The interventionists taught study participants the COPE (Creativity, Optimism, Planning, Expert Advice) model of problem solving and guided them through the application of this model in their caregiver role. They also receive tailored stroke education, specific to their needs through the RESCUE website.
Arm/Group | Standard Care Group | Intervention Group
Number analyzed (Participants) | 86 | 70
score on a scale | 15.0 (6.5) | 10.2 (5.4)
Statistical Analysis 1: Comparison: Standard Care Group vs Intervention Group; Test type: Superiority; p = 0.001, Mixed Models Analysis — a priori <0.05 threshold; Slope = -5.06, Standard Error of Mean 1.48 — Group X Time Interaction

2. Primary Outcome: Change in Caregiver Depression at 21 Weeks
Description: as for outcome 1
Time Frame: 21 weeks after baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care Group | Intervention Group
Number analyzed (Participants) | 86 | 70
score on a scale | 14.3 (7.7) | 10.5 (6.0)
Statistical Analysis 1: Comparison: Standard Care Group vs Intervention Group; Test type: Superiority; p = 0.017, Mixed Models Analysis — a priori <0.05 threshold; Slope = -4.04, Standard Error of Mean 1.69 — Group X Time Interaction

3. Secondary Outcome: Change in Caregiver Burden-Zarit - 9 Weeks
Description: Changes in burden will be measured by the Zarit Burden Interview instrument. This 22 item instrument is scored on a 5-point Likert scale, ranging from 0 (Never) to 4 (Nearly Always). The minimum value is 0 and the maximum score is 88. Higher scores indicate higher burden.
Time Frame: 9 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Problem Solving Intervention: Participants in the intervention group received an 8-week problem-solving session conducted over the phone by a trained interventionist. The intervention consists of four components: 1. Introduction to the RESCUE website and the problem-solving method; 2. Illustrative example on how to use the problem-solving approach and the RESCUE website to address caregiving problems; 3. Individualized practice exercise to develop a personalized problem-solving plan; and 4. Summary of the problem-solving method.
  RESCUE Problem Solving Intervention: The RESCUE Problem Solving Intervention: This is an education and support intervention for caregivers of Veterans with stroke. The interventionist taught study participants the COPE (Creativity, Optimism, Planning, Expert Advice) model of problem solving and guided them through the application of this model in their caregiver role. They also receive tailored stroke education, specific to their needs, based on the RESCUE website.
Arm/Group | Standard Care | Problem Solving Intervention
Number analyzed (Participants) | 86 | 70
score on a scale | 30.3 (5.9) | 24.5 (6.6)
Statistical Analysis 1: Comparison: Standard Care vs Problem Solving Intervention; Test type: Superiority; p = 0.017, Mixed Models Analysis — a priori of <0.05 threshold; Slope = -4.04, Standard Error of Mean 1.68 — Group X Time Interaction

4. Secondary Outcome: Change in Caregiver Burden-Zarit - 21 Weeks
Description: as for outcome 3
Time Frame: 21 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care | Problem Solving Intervention
Number analyzed (Participants) | 86 | 70
score on a scale | 30.8 (6.7) | 23.2 (7.0)
Statistical Analysis 1: Comparison: Standard Care vs Problem Solving Intervention; Test type: Superiority; p = 0.002, Mixed Models Analysis — a priori of <0.05 threshold; Slope = -5.66, Standard Error of Mean 1.84

5. Secondary Outcome: Change in Caregiver Self-Efficacy-Obtaining Respite - 9 Weeks
Description: Change in Self-Efficacy is measured by the Revised Scale for Caregiving Self-Efficacy- Obtaining Respite subscale. The subscale contains 5 items which asks caregivers to rate their level of confidence (from 0% to 100%) to ask for assistance. The subscale score is obtained by calculating the mean of the items, with a total score range of 0-100. Higher scores indicate higher self-efficacy. The subscale shows strong internal consistency and adequate test-retest reliability.
Time Frame: 9 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Intervention Group: Participants in the intervention group received an 8-week problem-solving session conducted over the phone by a trained interventionist. The intervention consists of four components: 1. Introduction to the RESCUE website and the problem-solving method; 2. Illustrative example on how to use the problem-solving approach and the RESCUE website to address caregiving problems; 3. Individualized practice exercise to develop a personalized problem-solving plan; and 4. Summary of the problem-solving method.
  The RESCUE Problem Solving Intervention: This is an education and support intervention for caregivers of Veterans with stroke. The interventionist taught study participants the COPE (Creativity, Optimism, Planning, Expert Advice) model of problem solving and guided them through the application of this model in their caregiver role. They also receive tailored stroke education, specific to their needs, based on the RESCUE website.
Arm/Group | Standard Care Group | Intervention Group
Number analyzed (Participants) | 86 | 70
score on a scale | 45.6 (18.2) | 54.2 (18.9)
Statistical Analysis 1: Comparison: Standard Care Group vs Intervention Group; Test type: Superiority; p = 0.152, Mixed Models Analysis — a priori of <0.05 threshold; Slope = 6.47, Standard Error of Mean 4.51 — Group x Time Interaction

6. Secondary Outcome: Change in Caregiver Self-Efficacy-Obtaining Respite - 21 Weeks
Description: as for outcome 5
Time Frame: 21 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care Group | Intervention Group
Number analyzed (Participants) | 86 | 70
score on a scale | 41.0 (17.3) | 57.2 (21.4)
Statistical Analysis 1: Comparison: Standard Care Group vs Intervention Group; Test type: Superiority; p = 0.008, Mixed Models Analysis — a priori of <0.05 threshold; Slope = 12.53, Standard Error of Mean 4.68 — Group x Time Interaction

7. Secondary Outcome: Changes in Caregiver Self-Efficacy- Controlling Upsetting Thoughts - 9 Weeks
Description: Measured by Revised Scale for Caregiver Self Efficacy - Controlling Upsetting Thoughts subscale (Steffen et al 2002). The subscale contains 5 items which ask caregivers to rate their level of confidence (from 0% to 100%) in their ability to control negative thoughts related to caregiving. The subscale score is obtained by calculating the mean of the items, with a total score range of 0-100. Higher scores indicate higher self-efficacy. The subscale shows strong internal consistency and adequate test-retest reliability.
Time Frame: 9 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care Group | Intervention Group
Number analyzed (Participants) | 86 | 70
score on a scale | 82.2 (9.0) | 84.8 (10.8)
Statistical Analysis 1: Comparison: Standard Care Group vs Intervention Group; Test type: Superiority; p = 0.812, Mixed Models Analysis — a priori of <0.05 threshold; Slope = 0.66, Standard Error of Mean 2.78 — Group X Time Interaction

8. Secondary Outcome: Changes in Caregiver Self-Efficacy- Controlling Upsetting Thoughts - 21 Weeks
Description: as for outcome 7
Time Frame: 21 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care Group | Intervention Group
Number analyzed (Participants) | 86 | 70
score on a scale | 79.9 (10.6) | 84.9 (10.6)
Statistical Analysis 1: Comparison: Standard Care Group vs Intervention Group; Test type: Superiority; p = 0.229, Mixed Models Analysis — a priori of <0.05 threshold; Slope = 3.64, Standard Error of Mean 3.02 — Group x Time Interaction

9. Secondary Outcome: Changes in Caregiver Self-Efficacy: Responding to Disruptive Behaviors - 9 Weeks
Description: Measured by Revised Scale for Caregiver Self Efficacy - Responding to Disruptive Behaviors subscale (Steffen et al 2002). The subscale contains 5 items which ask caregivers to rate their level of confidence (from 0% to 100%) in their ability to control negative thoughts related to caregiving. The subscale score is obtained by calculating the mean of the items, with a total score range of 0-100. Higher scores indicate higher self-efficacy. The subscale shows strong internal consistency and adequate test-retest reliability.
Time Frame: 9 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care Group | Intervention Group
Number analyzed (Participants) | 86 | 70
score on a scale | 81.2 (11.1) | 80.2 (11.1)
Statistical Analysis 1: Comparison: Standard Care Group vs Intervention Group; Test type: Superiority; p = 0.968, Mixed Models Analysis — a priori of <0.05 threshold; Slope = 0.21, Standard Error of Mean 5.25 — Group X Time Interaction

10. Secondary Outcome: Changes in Caregiver Self-Efficacy: Responding to Disruptive Behaviors - 21 Weeks
Description: as for outcome 9
Time Frame: 21 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care Group | Intervention Group
Number analyzed (Participants) | 86 | 70
score on a scale | 78.6 (9.2) | 86.6 (11.1)
Statistical Analysis 1: Comparison: Standard Care Group vs Intervention Group; Test type: Superiority; p = 0.196, Mixed Models Analysis — a priori of <0.05 threshold; Slope = 7.24, Standard Error of Mean 5.58 — Group X Time Interaction

11. Secondary Outcome: Change in Veteran's Functional Abilities- 9 Weeks
Description: Changes in Veteran functional abilities as measured by the Stroke Impact Scale-16 (SIS-16). The SIS-16 is a 16 item physical dimension instrument, developed as a brief standalone tool for measuring the physical aspects of stroke recovery. We modified this instrument to be administered to the caregiver about their evaluation of Veteran's functional ability. Scoring is based on a 5-point Likert scale, ranging from 16-80 points with 1 = an inability to complete the item & 5 = no difficulty experienced at all. Total Scores are transformed scores which have been standardized on a scale of 0-100 where higher scores indicate higher functional outcomes.
Time Frame: 9 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care Group | Intervention Group
Number analyzed (Participants) | 86 | 69
score on a scale | 43.8 (6.0) | 51.6 (8.3)
Statistical Analysis 1: Comparison: Standard Care Group vs Intervention Group; Test type: Superiority; p = 0.067, Mixed Models Analysis — a priori of <0.05 threshold; Slope = 3.46, Standard Error of Mean 1.89 — Group x Time Interaction

12. Secondary Outcome: Change in Veteran's Functional Abilities- 21 Weeks
Description: as for outcome 11
Time Frame: 21 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care Group | Intervention Group
Number analyzed (Participants) | 85 | 70
score on a scale | 43.3 (7.8) | 51.7 (9.3)
Statistical Analysis 1: Comparison: Standard Care Group vs Intervention Group; Test type: Superiority; p = 0.066, Mixed Models Analysis — a priori of <0.05 threshold; Slope = 3.98, Standard Error of Mean 2.16 — Group X Time Interaction

13. Secondary Outcome: Changes in Caregiver Health-Related Quality of Life - Physical Component Score - 9 Weeks
Description: Changes in health-related quality of life will be measured by the Rand 12-item Health Survey (VR-12). The VR12 items are scored on a 3-point or 5-point Likert scale. It consists of physical and emotional scales. Scores for each scale are calculated by using an algorithm and scores are standardized using a T-score metric with a mean of 50 and standard deviation of 10. Higher scores indicate better health-related quality of life. There is no composite or overall score for the VR-12.
Time Frame: 9 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Standard Care Group | Intervention Group
Number analyzed (Participants) | 86 | 70
T-score | 41.8 (6.1) | 42.8 (5.9)
Statistical Analysis 1: Comparison: Standard Care Group vs Intervention Group; Test type: Superiority; p = 0.225, Mixed Models Analysis — a priori of <0.05 threshold; Slope = 1.99, Standard Error of Mean 1.64 — Group X Time Interaction

14. Secondary Outcome: Changes in Caregiver Health-Related Quality of Life - Physical Component Score - 21 Weeks
Description: as for outcome 13
Time Frame: 21 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Standard Care Group | Intervention Group
Number analyzed (Participants) | 86 | 70
T-score | 40.3 (5.5) | 41.2 (5.9)
Statistical Analysis 1: Comparison: Standard Care Group vs Intervention Group; Test type: Superiority; p = 0.138, Mixed Models Analysis — a priori of <0.05 threshold; Slope = 1.93, Standard Error of Mean 1.30 — Group X Time Interaction

15. Secondary Outcome: Changes in Caregiver Health Related Quality of Life - Mental Health Component - 9 Weeks
Description: as for outcome 13
Time Frame: 9 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Groups:
- Intervention Group: Participants in the intervention group received an 8-week problem-solving session conducted over the phone by a trained interventionist. The intervention consists of four components: 1. Introduction to the RESCUE website and the problem-solving method; 2. Illustrative example on how to use the problem-solving approach and the RESCUE website to address caregiving problems; 3. Individualized practice exercise to develop a personalized problem-solving plan; and 4. Summary of the problem-solving method.
  The RESCUE Problem Solving Intervention: This is an education and support intervention for caregivers of Veterans with stroke. The interventionists taught study participants the COPE (Creativity, Optimism, Planning, Expert Advice) model of problem solving and guided them through the application of this model in their caregiver role. They also receive tailored stroke education, specific to their needs, based on the RESCUE website.
Arm/Group | Standard Care Group | Intervention Group
Number analyzed (Participants) | 86 | 70
T-score | 43.8 (6.7) | 49.9 (6.1)
Statistical Analysis 1: Comparison: Standard Care Group vs Intervention Group; Test type: Superiority; p = 0.002, Mixed Models Analysis — a priori of <0.05 threshold; Slope = 5.17, Standard Error of Mean 1.64 — Group x Time Interaction

16. Secondary Outcome: Changes in Caregiver Health Related Quality of Life - Mental Health Component - 21 Weeks
Description: as for outcome 13
Time Frame: 21 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Standard Care Group | Intervention Group
Number analyzed (Participants) | 86 | 70
T-score | 44.4 (6.5) | 48.4 (6.0)
Statistical Analysis 1: Comparison: Standard Care Group vs Intervention Group; Test type: Superiority; p = 0.052, Mixed Models Analysis — a priori of <0.05 threshold; Slope = 3.12, Standard Error of Mean 1.60 — Group X Time Interaction

17. Secondary Outcome: Social Problem-Solving Inventory-Revised Short Form (SPSI-R:S) -Change in Caregiver Problem Solving Abilities- Positive Problem Orientation (PPO) at 9 Weeks
Description: The Social Problem Solving Inventory Revised- Short Form (SPSI-R:S) is a 25-item, self-report instrument that evaluates characteristics of social problem solving, including problem solving orientation and problem solving performance. The SPSI-R:S consists of five subscores: positive problem orientation (PPO), negative problem orientation (NPO), rational problem solving style (RPS), impulsivity/carelessness style (ICS), and avoidance style (AS). Each sub-score contains five items that are scored on a five-point Likert-type rating scale, ranging from 0 (not at all true) to 4 (extremely true). Standardized scores range depending on the age of the person: Subscale PPO- 47-135; Subscale NPO= 74-162; Subscale RPS= 56-136; Subscale ICS= 73-162; Subscale AS= 76-157, Total SPSI= 29-140. Higher subscores on PPO and RPS, and lower subscores of NPO, ICS, and AS indicate good social problem solving.
Time Frame: 9 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care Group | Intervention Group
Number analyzed (Participants) | 86 | 70
score on a scale | 99.5 (10.3) | 98.0 (8.7)
Statistical Analysis 1: Comparison: Standard Care Group vs Intervention Group; Test type: Superiority; p = 0.981, Mixed Models Analysis — a priori of <0.05 threshold; Slope = -0.06, Standard Error of Mean 2.50 — Group X Time Interaction

18. Secondary Outcome: Social Problem-Solving Inventory-Revised Short Form (SPSI-R:S) -Change in Caregiver Problem Solving Abilities- Positive Problem Orientation (PPO) at 21 Weeks
Description: as for outcome 17
Time Frame: 21 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care Group | Intervention Group
Number analyzed (Participants) | 86 | 70
score on a scale | 98.2 (10.4) | 100.1 (10.7)
Statistical Analysis 1: Comparison: Standard Care Group vs Intervention Group; Test type: Superiority; p = 0.221, Mixed Models Analysis — a priori of <0.05 threshold; Slope = 3.29, Standard Error of Mean 2.68 — Group x Time Interaction

19. Secondary Outcome: Social Problem-Solving Inventory-Revised Short Form (SPSI-R:S) -Change in Caregiver Problem Solving Abilities- Negative Problem Orientation (NPO) at 9 Weeks
Description: as for outcome 17
Time Frame: 9 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care Group | Intervention Group
Number analyzed (Participants) | 86 | 70
score on a scale | 93.2 (7.6) | 92.1 (5.5)
Statistical Analysis 1: Comparison: Standard Care Group vs Intervention Group; Test type: Superiority; p = 0.159, Mixed Models Analysis — a priori of <0.05 threshold; Slope = -2.35, Standard Error of Mean 1.66 — Group x Time Interaction

20. Secondary Outcome: Social Problem-Solving Inventory-Revised Short Form (SPSI-R:S) -Change in Caregiver Problem Solving Abilities- Negative Problem Orientation (NPO) at 21 Weeks
Description: as for outcome 17
Time Frame: 21 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care Group | Intervention Group
Number analyzed (Participants) | 86 | 70
score on a scale | 92.5 (8.1) | 90.6 (7.7)
Statistical Analysis 1: Comparison: Standard Care Group vs Intervention Group; Test type: Superiority; p = 0.103, Mixed Models Analysis — a priori of <0.05 threshold; Slope = -3.13, Standard Error of Mean 1.91 — Group x Time Interaction

21. Secondary Outcome: Social Problem-Solving Inventory-Revised Short Form (SPSI-R:S) - Change in Caregiver Problem Solving Abilities- Rational Problem-Solving (RPS) at 9 Weeks
Description: as for outcome 17
Time Frame: 9 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care Group | Intervention Group
Number analyzed (Participants) | 86 | 70
score on a scale | 101.2 (9.5) | 105.0 (9.1)
Statistical Analysis 1: Comparison: Standard Care Group vs Intervention Group; Test type: Superiority; p = 0.247, Mixed Models Analysis — a priori of <0.05 threshold; Slope = 2.84, Standard Error of Mean 2.45 — Group x Time Interaction

22. Secondary Outcome: Social Problem-Solving Inventory-Revised Short Form (SPSI-R:S) -Change in Caregiver Problem Solving Abilities- Rational Problem-Solving (RPS) at 21 Weeks
Description: as for outcome 17
Time Frame: 21 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care Group | Intervention Group
Number analyzed (Participants) | 86 | 70
score on a scale | 100.5 (9.2) | 104.9 (10.2)
Statistical Analysis 1: Comparison: Standard Care Group vs Intervention Group; Test type: Superiority; p = 0.174, Mixed Models Analysis — a priori of <0.05 threshold; Slope = 3.43, Standard Error of Mean 2.52 — Group x Time Interaction

23. Secondary Outcome: Social Problem-Solving Inventory-Revised Short Form (SPSI-R:S) - Change in Caregiver Problem Solving Abilities- Impulsivity/Carelessness Style (ICS) at 9 Weeks
Description: as for outcome 17
Time Frame: 9 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care Group | Intervention Group
Number analyzed (Participants) | 86 | 70
score on a scale | 91.5 (9.1) | 92.4 (7.6)
Statistical Analysis 1: Comparison: Standard Care Group vs Intervention Group; Test type: Superiority; p = 0.408, Mixed Models Analysis — a priori of <0.05 threshold; Slope = 1.73, Standard Error of Mean 2.09 — Group x Time Interaction

24. Secondary Outcome: Social Problem-Solving Inventory-Revised Short Form (SPSI-R:S) - Change in Caregiver Problem Solving Abilities- Impulsivity/Carelessness Style (ICS) at 21 Weeks
Description: as for outcome 17
Time Frame: 21 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care Group | Intervention Group
Number analyzed (Participants) | 86 | 70
score on a scale | 91.7 (9.0) | 92.4 (7.5)
Statistical Analysis 1: Comparison: Standard Care Group vs Intervention Group; Test type: Superiority; p = 0.457, Mixed Models Analysis — a priori of <0.05 threshold; Slope = 1.53, Standard Error of Mean 2.06 — Group x Time Interaction

25. Secondary Outcome: Social Problem-Solving Inventory-Revised Short Form (SPSI-R:S) - Change in Caregiver Problem Solving Abilities- Avoidance Style (AS) at 9 Weeks
Description: as for outcome 17
Time Frame: 9 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care Group | Intervention Group
Number analyzed (Participants) | 86 | 70
score on a scale | 88.6 (7.8) | 87.7 (7.6)
Statistical Analysis 1: Comparison: Standard Care Group vs Intervention Group; Test type: Superiority; p = 0.187, Mixed Models Analysis — a priori of <0.05 threshold; Slope = -2.37, Standard Error of Mean 1.79 — Group x Time Interaction

26. Secondary Outcome: Social Problem-Solving Inventory-Revised Short Form (SPSI-R:S) -Change in Caregiver Problem Solving Abilities- Avoidance Style (AS) at 21 Weeks
Description: as for outcome 17
Time Frame: 21 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care Group | Intervention Group
Number analyzed (Participants) | 86 | 70
score on a scale | 87.4 (9.1) | 86.9 (7.9)
Statistical Analysis 1: Comparison: Standard Care Group vs Intervention Group; Test type: Superiority; p = 0.315, Mixed Models Analysis — a priori of <0.05 threshold; Slope = -2.00, Standard Error of Mean 1.99 — Group x Time Interaction

27. Secondary Outcome: Social Problem-Solving Inventory-Revised Short Form (SPSI-R:S) - Change in Caregiver Problem Solving Abilities- Problem Solving Total at 9 Weeks
Description: as for outcome 17
Time Frame: 9 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care Group | Intervention Group
Number analyzed (Participants) | 86 | 70
score on a scale | 107.7 (5.6) | 108.7 (5.7)
Statistical Analysis 1: Comparison: Standard Care Group vs Intervention Group; Test type: Superiority; p = 0.289, Mixed Models Analysis — a priori of <0.05 threshold; Slope = 1.49, Standard Error of Mean 1.41 — Group x Time Interaction

28. Secondary Outcome: Social Problem-Solving Inventory-Revised Short Form (SPSI-R:S) - Change in Caregiver Problem Solving Abilities- Problem Solving Total at 21 Weeks
Description: as for outcome 17
Time Frame: 21 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care Group | Intervention Group
Number analyzed (Participants) | 86 | 70
score on a scale | 107.5 (6.0) | 109.9 (6.4)
Statistical Analysis 1: Comparison: Standard Care Group vs Intervention Group; Test type: Superiority; p = 0.055, Mixed Models Analysis — a priori of <0.05 threshold; Slope = 2.92, Standard Error of Mean 1.52 — Group x Time Interaction

29. Other Pre Specified Outcome: Veteran's Healthcare Utilization - Number of Participants With Hospitalizations - 9 Weeks
Description: Veterans' Healthcare Utilization as measured by a survey developed for this study to record the number, dates, and the reasons for all healthcare visits (hospitalizations, ER, clinic visits) Veterans had during the course of the study. The survey consisted of ten questions with combined response choices including categorical (yes/no) and open responses (what was the reason for the visit). While the utilization variables are numerical, they are count variables with positive skew; the majority of values are 0, but with some values ranging from 1-4. Thus, we analyzed the variables as categorical (yes/no), using Chi-Square tests and providing values as frequencies.
Time Frame: 9 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Problem Solving Intervention: Participants in the intervention group received an 8-week problem-solving session conducted over the phone by a trained interventionist. The intervention consists of four components: 1. Introduction to the RESCUE website and the problem-solving method; 2. Illustrative example on how to use the problem-solving approach and the RESCUE website to address caregiving problems; 3. Individualized practice exercise to develop a personalized problem-solving plan; and 4. Summary of the problem-solving method.
  RESCUE Problem Solving Intervention: The RESCUE Problem Solving Intervention: This is an education and support intervention for caregivers of Veterans with stroke. The interventionists taught study participants the COPE (Creativity, Optimism, Planning, Expert Advice) model of problem solving and guided them through the application of this model in their caregiver role. They also receive tailored stroke education, specific to their needs, based on the RESCUE website.
Arm/Group | Standard Care | Problem Solving Intervention
Number analyzed (Participants) | 86 | 70
Participants | 9 | 14
Statistical Analysis 1: Comparison: Standard Care vs Problem Solving Intervention; Test type: Other; p = 0.095, Chi-squared

30. Other Pre Specified Outcome: Veteran's Healthcare Utilization - Number of Participants With Hospitalizations - 21 Weeks
Description: as for outcome 29
Time Frame: 21 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Problem Solving Intervention
Number analyzed (Participants) | 86 | 70
Participants | 11 | 11
Statistical Analysis 1: Comparison: Standard Care vs Problem Solving Intervention; Test type: Other; p = 0.6, Chi-squared

31. Other Pre Specified Outcome: Veteran's Healthcare Utilization - Number of Participants With Hospitalizations - Emergency Room Visits - 9 Weeks
Description: as for outcome 29
Time Frame: 9 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Problem Solving Intervention
Number analyzed (Participants) | 86 | 70
Participants | 28 | 33
Statistical Analysis 1: Comparison: Standard Care vs Problem Solving Intervention; Test type: Other; p = 0.063, Chi-squared

32. Other Pre Specified Outcome: Veteran's Healthcare Utilization - Number of Participants With Hospitalizations - Emergency Room Visits - 21 Weeks
Description: as for outcome 29
Time Frame: 21 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Problem Solving Intervention
Number analyzed (Participants) | 86 | 70
Participants | 30 | 25
Statistical Analysis 1: Comparison: Standard Care vs Problem Solving Intervention; Test type: Other; p = 0.9, Chi-squared

33. Other Pre Specified Outcome: Veteran's Healthcare Utilization - Number of Participants With Hospitalizations - Unplanned Primary Care Visits - 9 Weeks
Description: as for outcome 29
Time Frame: 9 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Problem Solving Intervention
Number analyzed (Participants) | 86 | 70
Participants | 10 | 14
Statistical Analysis 1: Comparison: Standard Care vs Problem Solving Intervention; Test type: Other; p = 0.15, Chi-squared

34. Other Pre Specified Outcome: Veteran's Healthcare Utilization - Number of Participants With Hospitalizations - Unplanned Primary Care Visits - 21 Weeks
Description: as for outcome 29
Time Frame: 21 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Problem Solving Intervention
Number analyzed (Participants) | 86 | 70
Participants | 13 | 18
Statistical Analysis 1: Comparison: Standard Care vs Problem Solving Intervention; Test type: Other; p = 0.11, Chi-squared

ADVERSE EVENTS:
Time Frame: from enrollment until end of post 2, up to 21 weeks.
Arm/Group | Standard Care Group | Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/105 | 0/105
Serious Adverse Events (participants affected / at risk) | 0/105 | 0/105
Other Adverse Events (participants affected / at risk) | 0/105 | 0/105

LIMITATIONS AND CAVEATS:
The study had no limitations or caveats.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-24): https://cdn.clinicaltrials.gov/large-docs/41/NCT03142841/Prot_SAP_001.pdf
  • Informed Consent Form (2023-08-28): https://cdn.clinicaltrials.gov/large-docs/41/NCT03142841/ICF_000.pdf